CLINICAL TRIAL: NCT05991778
Title: Bioelectrical Impedance Vector Analysis (BIVA) in Monitoring Hyperhydration and Polyneuromyopathy in Critically Ill Patients
Brief Title: Bioelectrical Impedance in Monitoring Hyperhydration and Polyneuromyopathy in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: KARIM-2022-BIVA; SGS09/LF/2022 (Other Grant/Funding Number: University of Ostrava)
Record Dates: First submitted 2023-07-27; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Distress Syndrome, Acute; Respiratory Insufficiency; Lung Ventilator; Hyperhydration; Hypoxemia; Chronic Obstructive Pulmonary Disease Exacerbation; Septic Shock
Keywords: Bioelectrical impedance; Hyperhydration; Critical care; Extracorporeal membrane oxygenation Mortality
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Water Intoxication; Hypoxia; Shock, Septic | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of Patients who Survived (S): The group is defined by the number of patients who survived.
  Interventions: Device: Bioelectrical impedance vector analysis (BIVA); Diagnostic Test: Blood and urine analysis; Diagnostic Test: cumulative water balance
- Group of Patients who Died (D): The group is defined by the number of patients who died.
  Interventions: Device: Bioelectrical impedance vector analysis (BIVA); Diagnostic Test: Blood and urine analysis; Diagnostic Test: cumulative water balance

INTERVENTIONS:
Device: Bioelectrical impedance vector analysis (BIVA) — BIVA is a simple, rapid, and noninvasive method, based on the principle that the flow of altering electrical current through a particular tissue differs depending on the content of water and electrolytes, used for monitoring hydratation and nutritional status in critically ill patients.
Diagnostic Test: Blood and urine analysis — For regular measurement in 2-3 terms, depending on the length of hospitalization (the first measurement took place within 48 hours of admission, followed one week after admission and the last before transport from the ICU): laboratory indicators of nutritional status will also be taken (albumin, prealbumin, creatinine), inflammation (C-reactive protein, presepsin) and 25-hydroxyvitamin D level.
Diagnostic Test: cumulative water balance — Cumulative balance is the sum of daily fluid balances during hospitalization.

SUMMARY:
This prospective, blinded observational clinical study was aimed to determine the effect of hyperhydration and muscle loss measured by Bioelectrical impedance vector analysis (BIVA) on mortality. The aim was to compare hydratation parameters measured by BIVA: OHY, Extracellular Water (ECW) / Total Body Wate (TBW) and quadrant, vector length, phase angle (PA) with cumulative fluid balance (CFB) recording (input-output) in their ability in predicting mortality as the abilities of the prognostic markers PA (BIVA), Acute Physiology and Chronic Health Evaluation II (APACHE II - score) and presepsin (serum Cluster of Differentiation (CD) 14-ST). The investigators also compared BIVA nutritional indicators (SMM, fat) with BMI and laboratory parameters (albumin, prealbumin and C-reactive protein (CRP) inflammation parameters) in the prediction of mortality. An important goal was to evaluate the usability of the BIVA method in critically ill patients on extracorporeal circulation, to compare the impedance data of the extracorporeal membrane oxygenation (ECMO) and non-ECMO groups.

DETAILED DESCRIPTION:
Hyperhydration has a detrimental effect on mortality risk and morbidity, increases the risk of acute kidney failure, the need of renal replacement therapy (RRT), worsens recovery of renal functions and worsens lung injury (ALI), infectious complications, and causes prolonged artificial pulmonary ventilation (APV), the length of stay on Intensive care unit (ICU), and impairs wound healing.

Real-time assessment of fluid status and management of fluid administration in critically ill patients is challenging. Echocardiography can rapidly identify hemodynamic phenotypes, but it is rather intermittent than continuous methods and requires experienced and trained staff. Semi-invasive methods, based on stroke volume monitoring as the area under the arterial curve and variability of stroke volume variation (SVV) evaluate intravascular volume. However, these methods lack information about the interstitial fluid, part of extracellular water (ECW), or intracellular fluid water (ICW). This problem is partially solved by transpulmonary thermodilution with extravascular lung water (EVLW) measurement and lung ultrasound. Calculating the cumulative balance (CBF) is imprecise, especially in the area of fluid output for insensible losses or third-space fluid losses. Even more imprecise is the clinical assessment of peripheral edema and blood flow. And gold standard deuterium dilution methods for total body water (TBW) are not usable in daily practice in the ICU settings.

In addition to hyperhydration, the rapid loss of muscle tissue in critically ill patients has a negative impact on the course of the disease. Polyneuromyopathy affects up to 40 % of critically ill patients, patients in a severe catabolic state with an activated systemic inflammatory response (SIRS), with corticosteroid therapy, and immobilized on long-term artificial lung ventilation are at risk. Monitoring lean body mass, especially skeletal muscle mass (SMM), is still difficult. Anthropometric measurements and ultrasound measurements of the quadriceps muscles are not ideal because they are time-consuming and require well-trained staff. Some laboratory parameters such as albumin are likely to be influenced by inflammation (CRP), and hydration. Dual-energy X-ray absorptiometers (DEXA) using two different wavelengths of low-intensity X-rays give a relatively accurate picture of bone mass and soft tissues (fat-free mass, active mass, fat). However, repeated X-ray examination in immobilized critically ill patients is not the method of choice.

Bioelectrical impedance vector analysis (BIVA) is a simple, rapid, and noninvasive bedside technique, based on the principle that the flow of altering electrical current through a particular tissue differs depending on the content of water and electrolytes. It is thus able to measure body composition as skeletal muscle mass (SMM), and body cell mass (BCM), including total body water and extracellular water. And with the use of 50 frequencies of bioimpedance spectroscopy (BIS), it is possible to distinguish TBW, ECW, and from their different intracellular water, because only electric current with a frequency higher than 100 Hertz (Hz) passes through the cell membrane. However, the technique cannot distinguish between intravascular and interstitial volumes in the extracellular compartment. According to a number of studies, the results of bioimpedance parameters of body composition are comparable to DEXA. However, BIA overestimates the representation of muscle. An important parameter is the phase angle (PA), which detects a time delay of the passage of current through the cell membrane, i.e., a phase shift between the sinusoidal voltage and current waveforms. PA reflects BCM and serves as an important prognostic factor, with a normal value of 4-15°.

Of the laboratory markers, presepsin (PSEP) has prognostic significance. Presepsin, soluble Cluster of differentiation 14 (sCD14), is a glycoprotein expressed in the membranes of monocytes and macrophages in response to pathogen-associated molecular patterns (PAMPs: lipopolysaccharide, peptidoglycan) part of the bacterial wall or to other damage to cells - damage-associated molecular patterns (DAMPs). An interesting finding is its prognostic role, i.e. higher values in non-surviving patients, evaluated by a number of studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory insufficiency, with the assumption of at least 7 days of artificial lung ventilation (medical, trauma, surgical patients)
* Primary acute respiratory distress syndrome (ARDS) (pulmonary involvement): pneumonia, inhalation trauma, chest trauma (lung contusion), aspiration
* Secondary ARDS (extrapulmonary): sepsis, shock states, acute pancreatitis, polytrauma, burns, non-cardiogenic shock, intoxication, TRALI (massive blood transfusion), drowning
* Patients with acute exacerbation of chronic obstructive pulmonary disease (COPD)

Exclusion Criteria:

* Patients with unfavorable prognosis
* APACHE II ≥30
* Metastatic malignancy
* Conditions after cardiopulmonary resuscitation (KPCR) before admission
* Cerebral edema
* Brain trauma
* Intracranial hypertension
* Liver cirrhosis
* A pre-existing neurodegenerative disease
* Patients with pacemakers, defibrillators, pregnancy (conditions contraindications to use of bio-electrical impedance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients admitted to 24 beds ICU of the University Hospital with the development of ARDS and the assumption of at least 7 days of artificial lung ventilation (medical, trauma, surgical patients) at the time of admission to the ICU.
  Informed consent was obtained from the person legally responsible for the patient.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Body Mass (physique) - Bioelectrical impedance analysis (BIA) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Bioelectrical impedance analysis (BIA) comparison of skeletal muscle mass, body fat and body water (expressed in %) in patients hospitalized in the ICU.
Body Mass (physique) - Phase Angle (PA) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Assessment of the Phase angle (expressed in degrees) as a part of BIA in patients hospitalized in the ICU.
Body Mass (physique) - BIVA vector analysis (Cole Cole graf) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Assessment of the BIVA vector analysis (Cole Cole graf, expressed as a optimal curve dependence of resistance on reactance always at a specific frequency, divided into quadrants) in patients hospitalized in the ICU.

SECONDARY OUTCOMES:
Indicators of nutritional status (albumin, prealbumin) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Assesment of indicators of nutritional status (albumin, prealbumin in g/l) in serum of patients admitted to Intensive Care Unit (ICU).
Indicator of inflammation (CRP) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Assesment of indicator of inflammation (C-reactive protein in mg/L) in serum of patients admitted to Intensive Care Unit (ICU).
Indicator of inflammation - presepsin (PSEP) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Assesment of indicator of inflammation measurements (presepsin in ng/L) in serum of patients admitted to Intensive Care Unit (ICU).

OTHER OUTCOMES:
Total body water (TBW) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Total body water measurements (in %) in patients admitted to Intensive Care Unit (ICU).
Extracellular water (ECW) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Extracellular water measurements (in %) in patients admitted to Intensive Care Unit (ICU).
Intracellular water (ICW) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Intracellular water measurements (in %) in patients admitted to Intensive Care Unit (ICU).
Overhydration (OHY) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Overhydration measurements (in %) in patients admitted to Intensive Care Unit (ICU).
Ratio ECW/TBW | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Ratio ECW/TBW measurements (in %) in patients admitted to Intensive Care Unit (ICU).
Active body mass index (ATH) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Active body mass index measurements (in kg/m2) in patients admitted to Intensive Care Unit (ICU).
Body mass index (BMI) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Body mass index measurements (in kg/m2) in patients admitted to Intensive Care Unit (ICU).
Body fat mass index (BFMI) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Body fat mass index measurements (in kg/m2) in patients admitted to Intensive Care Unit (ICU).
Fat-free mass index (FFMI) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Fat-free mass index measurements (in kg/m2) in patients admitted to Intensive Care Unit (ICU).
Skeletal muscle mass (SMM) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Skeletal muscle mass measurements (in kg) in patients admitted to Intensive Care Unit (ICU).
Body cell mass (BCM) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Body cell mass measurements (in kg) in patients admitted to Intensive Care Unit (ICU).
Basal metabolic rate (BMR) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Basal metabolic rate measurements (in kcal) in patients admitted to Intensive Care Unit (ICU).
Nutric index (NI) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Nutric index measurements (in %) in patients admitted to Intensive Care Unit (ICU).
Prediction marker (PM) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Prediction marker measurements in patients admitted to Intensive Care Unit (ICU). The mark value under 0,75 indicates normal condition, value over 0,86 means critical condition.
Indicators of nutritional status (creatinine) | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Indicators of nutritional status measurements (creatinine in µmol/L) in serum of patients admitted to Intensive Care Unit (ICU).
Level of 25-hydroxyvitamin D | The first within 48 hours of admission, the second one week after admission and third before transport from the ICU
  Level of 25-hydroxyvitamin D measurements (in nmol/L) in serum of patients admitted to Intensive Care Unit (ICU).
Cumulative fluid balance (CFB) | Every 24 hours until patient´s transport from the ICU
  Cumulative fluid balance daily measurements (in ml) in patients admitted to Intensive Care Unit (ICU).
Measurement of energy income | Every 24 hours until patient´s transport from the ICU
  Measurement of daily energy income (in kcals) in patients admitted to Intensive Care Unit (ICU).
Measurement of protein income | Every 24 hours until patient´s transport from the ICU
  Measurement of daily protein income (in g) in patients admitted to Intensive Care Unit (ICU).
Assessment of the presence of delirium (CAM-ICU test) | Every 24 hours until patient´s transport from the ICU
  The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) is a simple and short test that enables continuous monitoring of the patients in conditions of ICU (measured as positive/negative).

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Káňová, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Vincent JL. Fluid management in the critically ill. Kidney Int. 2019 Jul;96(1):52-57. doi: 10.1016/j.kint.2018.11.047. Epub 2019 Mar 4. PMID 30926137
- [Background] Payen D, de Pont AC, Sakr Y, Spies C, Reinhart K, Vincent JL; Sepsis Occurrence in Acutely Ill Patients (SOAP) Investigators. A positive fluid balance is associated with a worse outcome in patients with acute renal failure. Crit Care. 2008;12(3):R74. doi: 10.1186/cc6916. Epub 2008 Jun 4. PMID 18533029
- [Background] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lee J, Lo S, McArthur C, McGuiness S, Norton R, Myburgh J, Scheinkestel C, Su S. An observational study fluid balance and patient outcomes in the Randomized Evaluation of Normal vs. Augmented Level of Replacement Therapy trial. Crit Care Med. 2012 Jun;40(6):1753-60. doi: 10.1097/CCM.0b013e318246b9c6. PMID 22610181
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Wang N, Jiang L, Zhu B, Wen Y, Xi XM; Beijing Acute Kidney Injury Trial (BAKIT) Workgroup. Fluid balance and mortality in critically ill patients with acute kidney injury: a multicenter prospective epidemiological study. Crit Care. 2015 Oct 23;19:371. doi: 10.1186/s13054-015-1085-4. PMID 26494153
- [Background] Malbrain MLNG, Langer T, Annane D, Gattinoni L, Elbers P, Hahn RG, De Laet I, Minini A, Wong A, Ince C, Muckart D, Mythen M, Caironi P, Van Regenmortel N. Intravenous fluid therapy in the perioperative and critical care setting: Executive summary of the International Fluid Academy (IFA). Ann Intensive Care. 2020 May 24;10(1):64. doi: 10.1186/s13613-020-00679-3. PMID 32449147
- [Background] Nunes TS, Ladeira RT, Bafi AT, de Azevedo LC, Machado FR, Freitas FG. Duration of hemodynamic effects of crystalloids in patients with circulatory shock after initial resuscitation. Ann Intensive Care. 2014 Aug 1;4:25. doi: 10.1186/s13613-014-0025-9. eCollection 2014. PMID 25593742
- [Background] Magder S. Volume and its relationship to cardiac output and venous return. Crit Care. 2016 Sep 10;20(1):271. doi: 10.1186/s13054-016-1438-7. PMID 27613307
- [Background] Messmer AS, Zingg C, Muller M, Gerber JL, Schefold JC, Pfortmueller CA. Fluid Overload and Mortality in Adult Critical Care Patients-A Systematic Review and Meta-Analysis of Observational Studies. Crit Care Med. 2020 Dec;48(12):1862-1870. doi: 10.1097/CCM.0000000000004617. PMID 33009098
- [Background] Silversides JA, Perner A, Malbrain MLNG. Liberal versus restrictive fluid therapy in critically ill patients. Intensive Care Med. 2019 Oct;45(10):1440-1442. doi: 10.1007/s00134-019-05713-y. Epub 2019 Aug 9. No abstract available. PMID 31399779
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Jones SL, Tanaka A, Eastwood GM, Young H, Peck L, Bellomo R, Martensson J. Bioelectrical impedance vector analysis in critically ill patients: a prospective, clinician-blinded investigation. Crit Care. 2015 Aug 12;19(1):290. doi: 10.1186/s13054-015-1009-3. PMID 26260579
- [Background] De Backer D, Aissaoui N, Cecconi M, Chew MS, Denault A, Hajjar L, Hernandez G, Messina A, Myatra SN, Ostermann M, Pinsky MR, Teboul JL, Vignon P, Vincent JL, Monnet X. How can assessing hemodynamics help to assess volume status? Intensive Care Med. 2022 Oct;48(10):1482-1494. doi: 10.1007/s00134-022-06808-9. Epub 2022 Aug 10. PMID 35945344
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Perren A, Markmann M, Merlani G, Marone C, Merlani P. Fluid balance in critically ill patients. Should we really rely on it? Minerva Anestesiol. 2011 Aug;77(8):802-11. PMID 21730928
- [Background] Preiser JC, Ichai C, Orban JC, Groeneveld AB. Metabolic response to the stress of critical illness. Br J Anaesth. 2014 Dec;113(6):945-54. doi: 10.1093/bja/aeu187. Epub 2014 Jun 26. PMID 24970271
- [Background] Kanova M, Kohout P. Molecular Mechanisms Underlying Intensive Care Unit-Acquired Weakness and Sarcopenia. Int J Mol Sci. 2022 Jul 29;23(15):8396. doi: 10.3390/ijms23158396. PMID 35955530
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Binkovitz LA, Henwood MJ. Pediatric DXA: technique and interpretation. Pediatr Radiol. 2007 Jan;37(1):21-31. doi: 10.1007/s00247-006-0153-y. Epub 2006 May 20. PMID 16715219
- [Background] Abramowitz MK, Hall CB, Amodu A, Sharma D, Androga L, Hawkins M. Muscle mass, BMI, and mortality among adults in the United States: A population-based cohort study. PLoS One. 2018 Apr 11;13(4):e0194697. doi: 10.1371/journal.pone.0194697. eCollection 2018. PMID 29641540
- [Background] Malbrain ML, Huygh J, Dabrowski W, De Waele JJ, Staelens A, Wauters J. The use of bio-electrical impedance analysis (BIA) to guide fluid management, resuscitation and deresuscitation in critically ill patients: a bench-to-bedside review. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):381-91. doi: 10.5603/AIT.2014.0061. PMID 25432557
- [Background] Basso F, Berdin G, Virzi GM, Mason G, Piccinni P, Day S, Cruz DN, Wjewodzka M, Giuliani A, Brendolan A, Ronco C. Fluid management in the intensive care unit: bioelectrical impedance vector analysis as a tool to assess hydration status and optimal fluid balance in critically ill patients. Blood Purif. 2013;36(3-4):192-9. doi: 10.1159/000356366. Epub 2013 Dec 20. PMID 24496190
- [Background] Moissl UM, Wabel P, Chamney PW, Bosaeus I, Levin NW, Bosy-Westphal A, Korth O, Muller MJ, Ellegard L, Malmros V, Kaitwatcharachai C, Kuhlmann MK, Zhu F, Fuller NJ. Body fluid volume determination via body composition spectroscopy in health and disease. Physiol Meas. 2006 Sep;27(9):921-33. doi: 10.1088/0967-3334/27/9/012. Epub 2006 Jul 25. PMID 16868355
- [Background] Khalil SF, Mohktar MS, Ibrahim F. The theory and fundamentals of bioimpedance analysis in clinical status monitoring and diagnosis of diseases. Sensors (Basel). 2014 Jun 19;14(6):10895-928. doi: 10.3390/s140610895. PMID 24949644
- [Background] Fujimoto K, Inage K, Eguchi Y, Orita S, Suzuki M, Kubota G, Sainoh T, Sato J, Shiga Y, Abe K, Kanamoto H, Inoue M, Kinoshita H, Norimoto M, Umimura T, Koda M, Furuya T, Akazawa T, Toyoguchi T, Terakado A, Takahashi K, Ohtori S. Use of Bioelectrical Impedance Analysis for the Measurement of Appendicular Skeletal Muscle Mass/Whole Fat Mass and Its Relevance in Assessing Osteoporosis among Patients with Low Back Pain: A Comparative Analysis Using Dual X-ray Absorptiometry. Asian Spine J. 2018 Oct;12(5):839-845. doi: 10.31616/asj.2018.12.5.839. Epub 2018 Sep 10. PMID 30213166
- [Background] Kushner RF, Schoeller DA, Fjeld CR, Danford L. Is the impedance index (ht2/R) significant in predicting total body water? Am J Clin Nutr. 1992 Nov;56(5):835-9. doi: 10.1093/ajcn/56.5.835. PMID 1415001
- [Background] Lukaski HC, Hall CB, Siders WA. Assessment of change in hydration in women during pregnancy and postpartum with bioelectrical impedance vectors. Nutrition. 2007 Jul-Aug;23(7-8):543-50. doi: 10.1016/j.nut.2007.05.001. Epub 2007 Jun 14. PMID 17570642
- [Background] Cheng KY, Chow SK, Hung VW, Wong CH, Wong RM, Tsang CS, Kwok T, Cheung WH. Diagnosis of sarcopenia by evaluating skeletal muscle mass by adjusted bioimpedance analysis validated with dual-energy X-ray absorptiometry. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):2163-2173. doi: 10.1002/jcsm.12825. Epub 2021 Oct 4. PMID 34609065
- [Background] Dzator S, Weerasekara I, Shields M, Haslam R, James D. Agreement Between Dual-Energy X-ray Absorptiometry and Bioelectric Impedance Analysis for Assessing Body Composition in Athletes: A Systematic Review and Meta-Analysis. Clin J Sport Med. 2023 Sep 1;33(5):557-568. doi: 10.1097/JSM.0000000000001136. Epub 2023 Feb 28. PMID 36853902
- [Background] Baumgartner RN, Chumlea WC, Roche AF. Bioelectric impedance phase angle and body composition. Am J Clin Nutr. 1988 Jul;48(1):16-23. doi: 10.1093/ajcn/48.1.16. PMID 3389323
- [Background] Gupta D, Lammersfeld CA, Burrows JL, Dahlk SL, Vashi PG, Grutsch JF, Hoffman S, Lis CG. Bioelectrical impedance phase angle in clinical practice: implications for prognosis in advanced colorectal cancer. Am J Clin Nutr. 2004 Dec;80(6):1634-8. doi: 10.1093/ajcn/80.6.1634. PMID 15585779
- [Background] Di Vincenzo O, Marra M, Di Gregorio A, Pasanisi F, Scalfi L. Bioelectrical impedance analysis (BIA) -derived phase angle in sarcopenia: A systematic review. Clin Nutr. 2021 May;40(5):3052-3061. doi: 10.1016/j.clnu.2020.10.048. Epub 2020 Nov 1. PMID 33183880
- [Background] Kyle UG, Soundar EP, Genton L, Pichard C. Can phase angle determined by bioelectrical impedance analysis assess nutritional risk? A comparison between healthy and hospitalized subjects. Clin Nutr. 2012 Dec;31(6):875-81. doi: 10.1016/j.clnu.2012.04.002. Epub 2012 May 4. PMID 22560739
- [Background] Gupta D, Lis CG, Dahlk SL, Vashi PG, Grutsch JF, Lammersfeld CA. Bioelectrical impedance phase angle as a prognostic indicator in advanced pancreatic cancer. Br J Nutr. 2004 Dec;92(6):957-62. doi: 10.1079/bjn20041292. PMID 15613258
- [Background] Gupta D, Lammersfeld CA, Vashi PG, King J, Dahlk SL, Grutsch JF, Lis CG. Bioelectrical impedance phase angle as a prognostic indicator in breast cancer. BMC Cancer. 2008 Aug 27;8:249. doi: 10.1186/1471-2407-8-249. PMID 18727837
- [Background] Kanova M, Dobias R, Liszkova K, Frelich M, Jecminkova R, Kula R. [Presepsin in the diagnostics of sepsis]. Vnitr Lek. 2019 Summer;65(7-8):497-505. Czech. PMID 31487993
- [Background] Behnes M, Bertsch T, Lepiorz D, Lang S, Trinkmann F, Brueckmann M, Borggrefe M, Hoffmann U. Diagnostic and prognostic utility of soluble CD 14 subtype (presepsin) for severe sepsis and septic shock during the first week of intensive care treatment. Crit Care. 2014 Sep 5;18(5):507. doi: 10.1186/s13054-014-0507-z. PMID 25190134
- [Background] Chamney PW, Wabel P, Moissl UM, Muller MJ, Bosy-Westphal A, Korth O, Fuller NJ. A whole-body model to distinguish excess fluid from the hydration of major body tissues. Am J Clin Nutr. 2007 Jan;85(1):80-9. doi: 10.1093/ajcn/85.1.80. PMID 17209181
- [Background] Piccoli A, Codognotto M, Piasentin P, Naso A. Combined evaluation of nutrition and hydration in dialysis patients with bioelectrical impedance vector analysis (BIVA). Clin Nutr. 2014 Aug;33(4):673-7. doi: 10.1016/j.clnu.2013.08.007. Epub 2013 Aug 31. PMID 24055204
- [Background] Peacock Iv WF. Use of bioimpedance vector analysis in critically ill and cardiorenal patients. Contrib Nephrol. 2010;165:226-235. doi: 10.1159/000313762. Epub 2010 Apr 20. PMID 20427973
- [Background] Piccoli A. Bioelectric impedance measurement for fluid status assessment. Contrib Nephrol. 2010;164:143-152. doi: 10.1159/000313727. Epub 2010 Apr 20. PMID 20428000
- [Background] Chen H, Wu B, Gong D, Liu Z. Fluid overload at start of continuous renal replacement therapy is associated with poorer clinical condition and outcome: a prospective observational study on the combined use of bioimpedance vector analysis and serum N-terminal pro-B-type natriuretic peptide measurement. Crit Care. 2015 Apr 2;19(1):135. doi: 10.1186/s13054-015-0871-3. PMID 25879573
- [Background] Finn PJ, Plank LD, Clark MA, Connolly AB, Hill GL. Progressive cellular dehydration and proteolysis in critically ill patients. Lancet. 1996 Mar 9;347(9002):654-6. doi: 10.1016/s0140-6736(96)91204-0. PMID 8596380
- [Background] Plank LD, Monk DN, Woollard GA, Hill GL. Evaluation of multifrequency bioimpedance spectroscopy for measurement of the extracellular water space in critically ill patients. Appl Radiat Isot. 1998 May-Jun;49(5-6):481-3. doi: 10.1016/s0969-8043(97)00060-2. PMID 9569521
- [Background] Dewitte A, Carles P, Joannes-Boyau O, Fleureau C, Roze H, Combe C, Ouattara A. Bioelectrical impedance spectroscopy to estimate fluid balance in critically ill patients. J Clin Monit Comput. 2016 Apr;30(2):227-33. doi: 10.1007/s10877-015-9706-7. Epub 2015 May 29. PMID 26018457
- [Background] Samoni S, Vigo V, Resendiz LI, Villa G, De Rosa S, Nalesso F, Ferrari F, Meola M, Brendolan A, Malacarne P, Forfori F, Bonato R, Donadio C, Ronco C. Impact of hyperhydration on the mortality risk in critically ill patients admitted in intensive care units: comparison between bioelectrical impedance vector analysis and cumulative fluid balance recording. Crit Care. 2016 Apr 8;20:95. doi: 10.1186/s13054-016-1269-6. PMID 27060079
- [Background] Yang SF, Tseng CM, Liu IF, Tsai SH, Kuo WS, Tsao TP. Clinical Significance of Bioimpedance Spectroscopy in Critically Ill Patients. J Intensive Care Med. 2019 Jun;34(6):495-502. doi: 10.1177/0885066617702591. Epub 2017 Apr 4. PMID 28372500
- [Background] Wang Y, Gu Z. Effect of bioimpedance-defined overhydration parameters on mortality and cardiovascular events in patients undergoing dialysis: a systematic review and meta-analysis. J Int Med Res. 2021 Sep;49(9):3000605211031063. doi: 10.1177/03000605211031063. PMID 34496645
- [Background] Park CS, Lee SE, Cho HJ, Kim YJ, Kang HJ, Oh BH, Lee HY. Body fluid status assessment by bio-impedance analysis in patients presenting to the emergency department with dyspnea. Korean J Intern Med. 2018 Sep;33(5):911-921. doi: 10.3904/kjim.2016.358. Epub 2017 Dec 18. PMID 29241303
- [Background] Yamazoe M, Mizuno A, Niwa K, Isobe M. Edema index measured by bioelectrical impedance analysis as a predictor of fluid reduction needed to remove clinical congestion in acute heart failure. Int J Cardiol. 2015 Dec 15;201:190-2. doi: 10.1016/j.ijcard.2015.07.086. Epub 2015 Jul 30. No abstract available. PMID 26298378
- [Background] Parrinello G, Paterna S, Di Pasquale P, Torres D, Fatta A, Mezzero M, Scaglione R, Licata G. The usefulness of bioelectrical impedance analysis in differentiating dyspnea due to decompensated heart failure. J Card Fail. 2008 Oct;14(8):676-86. doi: 10.1016/j.cardfail.2008.04.005. Epub 2008 Jun 6. PMID 18926440
- [Background] Genot N, Mewton N, Bresson D, Zouaghi O, Francois L, Delwarde B, Kirkorian G, Bonnefoy-Cudraz E. Bioelectrical impedance analysis for heart failure diagnosis in the ED. Am J Emerg Med. 2015 Aug;33(8):1025-9. doi: 10.1016/j.ajem.2015.04.021. Epub 2015 Apr 20. PMID 25959843
- [Background] Gil Martinez P, Mesado Martinez D, Curbelo Garcia J, Cadinanos Loidi J. Amino-terminal pro-B-type natriuretic peptide, inferior vena cava ultrasound, and biolectrical impedance analysis for the diagnosis of acute decompensated CHF. Am J Emerg Med. 2016 Sep;34(9):1817-22. doi: 10.1016/j.ajem.2016.06.043. Epub 2016 Jun 14. PMID 27396536
- [Background] Di Somma S, Lalle I, Magrini L, Russo V, Navarin S, Castello L, Avanzi GC, Di Stasio E, Maisel A. Additive diagnostic and prognostic value of bioelectrical impedance vector analysis (BIVA) to brain natriuretic peptide 'grey-zone' in patients with acute heart failure in the emergency department. Eur Heart J Acute Cardiovasc Care. 2014 Jun;3(2):167-75. doi: 10.1177/2048872614521756. Epub 2014 Jan 29. PMID 24477201
- [Background] Dabrowski W, Kotlinska-Hasiec E, Schneditz D, Zaluska W, Rzecki Z, De Keulenaer B, Malbrain ML. Continuous veno-venous hemofiltration to adjust fluid volume excess in septic shock patients reduces intra-abdominal pressure. Clin Nephrol. 2014 Jul;82(1):41-50. doi: 10.5414/CN108015. PMID 24887300
- [Background] Malbrain ML, Marik PE, Witters I, Cordemans C, Kirkpatrick AW, Roberts DJ, Van Regenmortel N. Fluid overload, de-resuscitation, and outcomes in critically ill or injured patients: a systematic review with suggestions for clinical practice. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):361-80. doi: 10.5603/AIT.2014.0060. PMID 25432556
- [Background] Slobod D, Yao H, Mardini J, Natkaniec J, Correa JA, Jayaraman D, Weber CL. Bioimpedance-measured volume overload predicts longer duration of mechanical ventilation in intensive care unit patients. Can J Anaesth. 2019 Dec;66(12):1458-1463. doi: 10.1007/s12630-019-01450-4. Epub 2019 Jul 23. PMID 31338808
- [Background] Colin-Ramirez E, Castillo-Martinez L, Orea-Tejeda A, Asensio Lafuente E, Torres Villanueva F, Rebollar Gonzalez V, Narvaez David R, Dorantes Garcia J. Body composition and echocardiographic abnormalities associated to anemia and volume overload in heart failure patients. Clin Nutr. 2006 Oct;25(5):746-57. doi: 10.1016/j.clnu.2006.01.009. Epub 2006 May 15. PMID 16698139
- [Background] Gulatava N, Tabagari N, Tabagari S. BIOELECTRICAL IMPENDANCE ANALYSIS OF BODY COMPOSITION IN PATIENTS WITH CHRONIC HEART FAILURE. Georgian Med News. 2021 Jun;(315):94-98. PMID 34365432
- [Background] Thibault R, Makhlouf AM, Mulliez A, Cristina Gonzalez M, Kekstas G, Kozjek NR, Preiser JC, Rozalen IC, Dadet S, Krznaric Z, Kupczyk K, Tamion F, Cano N, Pichard C; Phase Angle Project Investigators. Fat-free mass at admission predicts 28-day mortality in intensive care unit patients: the international prospective observational study Phase Angle Project. Intensive Care Med. 2016 Sep;42(9):1445-53. doi: 10.1007/s00134-016-4468-3. Epub 2016 Aug 11. PMID 27515162
- [Background] Lukaski HC, Kyle UG, Kondrup J. Assessment of adult malnutrition and prognosis with bioelectrical impedance analysis: phase angle and impedance ratio. Curr Opin Clin Nutr Metab Care. 2017 Sep;20(5):330-339. doi: 10.1097/MCO.0000000000000387. PMID 28548972
- [Background] Tanaka S, Ando K, Kobayashi K, Seki T, Hamada T, Machino M, Ota K, Morozumi M, Kanbara S, Ito S, Ishiguro N, Hasegawa Y, Imagama S. Low Bioelectrical Impedance Phase Angle Is a Significant Risk Factor for Frailty. Biomed Res Int. 2019 Jun 10;2019:6283153. doi: 10.1155/2019/6283153. eCollection 2019. PMID 31281842
- [Background] Varan HD, Bolayir B, Kara O, Arik G, Kizilarslanoglu MC, Kilic MK, Sumer F, Kuyumcu ME, Yesil Y, Yavuz BB, Halil M, Cankurtaran M. Phase angle assessment by bioelectrical impedance analysis and its predictive value for malnutrition risk in hospitalized geriatric patients. Aging Clin Exp Res. 2016 Dec;28(6):1121-1126. doi: 10.1007/s40520-015-0528-8. Epub 2016 Jan 19. PMID 26786583
- [Background] Looijaard WGPM, Stapel SN, Dekker IM, Rusticus H, Remmelzwaal S, Girbes ARJ, Weijs PJM, Oudemans-van Straaten HM. Identifying critically ill patients with low muscle mass: Agreement between bioelectrical impedance analysis and computed tomography. Clin Nutr. 2020 Jun;39(6):1809-1817. doi: 10.1016/j.clnu.2019.07.020. Epub 2019 Aug 10. PMID 31492456
- [Background] Moonen HPFX, Van Zanten ARH. Bioelectric impedance analysis for body composition measurement and other potential clinical applications in critical illness. Curr Opin Crit Care. 2021 Aug 1;27(4):344-353. doi: 10.1097/MCC.0000000000000840. PMID 33967207
- [Background] Latronico N, Bolton CF. Critical illness polyneuropathy and myopathy: a major cause of muscle weakness and paralysis. Lancet Neurol. 2011 Oct;10(10):931-41. doi: 10.1016/S1474-4422(11)70178-8. PMID 21939902
- [Background] Rousseau AF, Prescott HC, Brett SJ, Weiss B, Azoulay E, Creteur J, Latronico N, Hough CL, Weber-Carstens S, Vincent JL, Preiser JC. Long-term outcomes after critical illness: recent insights. Crit Care. 2021 Mar 17;25(1):108. doi: 10.1186/s13054-021-03535-3. PMID 33731201